CLINICAL TRIAL: NCT05117242
Title: A Phase 2, Multicenter, Randomized, Open-Label Trial of GEN1046 as Monotherapy and in Combination Pembrolizumab Therapy in Subjects With Relapsed/Refractory Metastatic Non-Small Cell Lung Cancer After Treatment With Standard of Care Therapy With an Immune Checkpoint Inhibitor
Brief Title: Safety and Efficacy Study of GEN1046 as a Single Agent or in Combination With Pembrolizumab for Treatment of Recurrent (Non-small Cell) Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-04; 2021-001928-17 (EudraCT Number); 1004314 (Other: IRAS ID; UK Research Summaries Database); NL-OMON54259 (Registry Identifier: CCMO (The Netherlands)); 2024-513770-22-00 (Other: EU Trial (CTIS) Number); RECF-005102 (Registry Identifier: National Institute of Cancer France); 15582 (Registry Identifier: Portugal RNET)
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: DuoBody®; Bispecific antibody; PD-L1; 4-1BB
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Treatment with acasunlimab once every 21 days for the first 2 cycles and then every 42 days in subsequent cycles
  Interventions: Biological: Acasunlimab
- Arm B (Experimental): Treatment with acasunlimab + pembrolizumab once every 21 days
  Interventions: Biological: Acasunlimab; Biological: Pembrolizumab
- Arm C (Experimental): Treatment with acasunlimab + pembrolizumab once every 42 days
  Interventions: Biological: Acasunlimab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Acasunlimab — Acasunlimab will be administered intravenously (IV)
  Other Names: GEN1046; DuoBody®-PD-L1×4-1BB
Biological: Pembrolizumab — Pembrolizumab will be administered IV
  Other Names: KEYTRUDA®
  Arms: Arm B; Arm C

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy (how well the drug works) of acasunlimab (also known as GEN1046) when it is used alone (monotherapy) versus when it is combined with a cancer drug (pembrolizumab) for participants with relapsed/refractory (disease has returned after treatment or did not respond to treatment) non-small cell lung cancer (NSCLC; the most common type of lung cancer).

This trial has 2 parts. The purpose of the first part is to find out if the combination of acasunlimab and pembrolizumab is safe and to find out the best doses to use. The purpose of the second part is to give acasunlimab and pembrolizumab to more participants to evaluate efficacy. In the second part of the trial, participants will be randomized to participate in 1 of the 3 arms of the trial. Randomized means that the participant will be randomly assigned to a treatment arm based on chance; no one chooses their treatment arm.

Participants will receive either acasunlimab alone (100 followed by 500 mg into the vein) or acasunlimab with pembrolizumab (200 or 400 mg into the vein) once every 3 or 6 weeks, depending on which arm the participant is randomized into. All participants will receive active drug; no one will receive placebo.

Trial details include:

* The average trial duration for an individual participant will be about 10 months.
* The average treatment duration for an individual participant will be about 6 months.
* The visit frequency will be weekly at first and lessening over time until visits are only once every 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Have signed an informed consent form (ICF)
* Be at least 18 years of age.
* Have histologically or cytologically confirmed diagnosis of stage 4 NSCLC with at least 1 prior line of systemic therapy containing an anti-PD-1/PD-L1 mAb for metastatic disease
* Have a tumor PD-L1 expression result available prior to first treatment demonstrating PD-L1 expression in ≥1% of tumor cells as assessed by a central or local laboratory during screening.
* Have measurable disease per RECIST v1.1.
* Have Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
* Have life expectancy of at least 3 months.
* Have adequate organ and bone marrow function as defined in the protocol.

Key Exclusion Criteria:

* Documentation of known EGFR, KRAS, RET, ROS1, BRAF mutations, NTRK gene infusions, RET arrangement, ALK gene rearrangements, high-level MET amplification, or METex 14 skipping. Note: Subjects harboring such mutations, gene rearrangements or amplifications may be enrolled in the trial, if subjects have received prior approved targeted therapy for such mutations, the subject may still be eligible for this trial.
* Treatment with an anti-cancer agent within 28 days prior to acasunlimab administration.
* Any investigational agent (including investigational vaccines).
* Radiotherapy within 14 days prior to first dose of acasunlimab. Note: palliative radiotherapy will be allowed for local pain control under certain conditions.
* Chronic systemic immunosuppressive corticosteroid doses, ie, prednisone >10 mg daily or a cumulative dose >150 mg prednisone within 14 days before the first acasunlimab administration.
* Subject has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Subject has contraindications to the use of pembrolizumab per local prescribing information.
* Subject has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis (interstitial lung disease).
* Ongoing or active infection requiring intravenous treatment with anti-infective therapy or any ongoing systemic inflammatory condition requiring further diagnostic work-up or management during screening.
* Symptomatic congestive heart failure (grade III or IV as classified by the New York Heart Association), unstable angina pectoris, or cardiac arrhythmia.
* Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg, despite optimal medical management.
* Ongoing or recent (within 6 months) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for irAEs.
* Subject has a known history of any of the following:

  1. Grade 3 or higher irAEs that led to treatment discontinuation of a prior immunotherapy treatment.
  2. Myositis, Guillain-Barré syndrome, or myasthenia gravis of any grade.
  3. Liver disease (eg, alcoholic hepatitis or non-alcoholic steatohepatitis, drug-related or autoimmune hepatitis, or evidence of hepatic cirrhosis).
  4. Organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of acasunlimab.
  5. Grade 3 or higher allergic reactions to monoclonal antibody therapy as well as known or suspected allergy or intolerance to any agent given in the course of this trial.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From first treatment to approximately 27 weeks after last subject's first dose
  ORR will be measured as the proportion of subjects with a confirmed response of complete response (CR) or partial response (PR) as per RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | From onset date of response until disease progression/death/lost to follow-up/start of new anticancer therapy or withdrawal of consent, whichever occurs first (an expected average of 6 months)
  DOR will be measured as the time from initial onset of CR or PR to first radiographic progression as per RECIST v. 1.1 or death from any cause, whichever occurs first.
Time to response (TTR) | From first treatment to date of onset of initial response (CR or PR) as per RECIST v.1.1 (an expected average of 6 months)
  TTR will be measured as the time from first treatment to onset of initial response (CR or PR) as per RECIST v.1.1
Progression-free survival (PFS) | From first treatment to first documented progression or death due to any cause (an expected average of 6 months)
  PFS will be measured from date of first treatment until date of radiographic progression as per RECIST v.1.1 or until death from any cause, whichever occurs first
Overall survival (OS) | From first treatment to date of death (assessed up to 3 years after the last participant's first dose in the trial)
  Defined as time to death from of any cause
Incidence and severity of adverse events (AEs) and laboratory abnormalities | Throughout the trial until end of safety follow-up period (60 days or 90 days after last dose)
  Incidence of treatment-emergent AEs as assessed by CTCAE v5.0. Laboratory parameters graded by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (40):
- United States (6):
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Florida Cancer Specialists - FCS South, Fort Myers, Florida
  - Florida Cancer Center, St. Petersburg, Florida
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan CHCWM P.C., Grand Rapids, Michigan
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (7):
  - Institut Bergonie, Bordeaux
  - Hopital Morvan CHU de Brest, Brest
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - Hopital dInstruction Des Armees Begin, Saint-Mandé
  - Institut de Cancerologie Strasbourg Europe (ICANS), Strasbourg
  - Hôpital Foch, Suresnes
  - Gustave Roussy, Villejuif
- Germany (4):
  - Med.Hochschule Hannover Klinik für Pneumologie, Hanover
  - Universitatsklinik Giessen und Marburg Standort Giessen, Hessen
  - LKI Lungenfachklinik Immenhausen, Immenhausen
  - Department of Internal Medicine II, Regensburg
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico G Rodolico San Marco, Catania
  - IRCCS Istituto Europeo di Oncologia, Milan
  - UOC Oncoematologia AOU L.Vanvitelli, Napoli
  - La Maddalena SPA, Palermo
  - IFO Regina Elena, Roma
- Netherlands (4):
  - Netherlands Cancer Institute, Amsterdam
  - VU University Medical Center, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC, Rotterdam
- Poland (2):
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Portugal (2):
  - Centro Clinico Champalimaud, Lisbon
  - Centro Hospitalar Universitário do Porto - Hospital de Santo Antonio, Porto
- Spain (8):
  - Hospital Universitari Vall dHebron, Barcelona
  - Clinica Universidad de Navarra CUN, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- United Kingdom (2):
  - Cheltenham General Hospital, Cheltenham
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No